CLINICAL TRIAL: NCT07058311
Title: Evaluation of the Effects of Physiotherapy and Rehabilitation Interventions in Patients With Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Miraç Sezer, lecturer, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-1166
Record Dates: First submitted 2025-05-09; First posted 2025-07-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Bruxism; Physiotherapy; Exercise; Manual Theapy; Pain
Keywords: Bruxism; Manual Therapy; Exercise; Ultrasonography; Electromyography; physiotherapy
MeSH Terms: conditions — Bruxism; Motor Activity; Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Thirty patients with bruxism were randomly divided into as Manual Therapy Group (15) and Home Exercise Group (15).
Who Masked: Participant, Outcomes Assessor
Masking Description: To ensure blinding, baseline and final outcome measurements were performed by researchers other than the physiotherapist performing manual therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy Group (Experimental): The term manual therapy includes a wide variety of detailed applications ranging from joint-oriented applications (joint mobilizations and/or manipulations) or soft tissue techniques (muscle stretching or trigger point therapy) to therapeutic exercises. Manual therapy in our study was used to restore normal temporomandibular joint range of motion, reduce local ischemia, stimulate proprioception, break fibrous adhesions, stimulate synovial fluid production and reduce pain.
  Interventions: Other: Manual Therapy
- Exercise Group (Experimental): Exercise therapy, one of the physical therapy applications, has an important place in the rehabilitation of musculoskeletal disorders. With this method, it is aimed to decrease inflammation, increase coordination of muscle activity, promote tissue repair and regeneration, relieve pain and restore normal function. In addition to the special exercises known as Rocabado exercises which are used in the treatment of temporomandibular joint, various studies have been performed in which mobilization, coordination, posture and relaxation exercises were used for the treatment of disorders related to the masticatory system and it has been emphasized that studies on this subject should be continued.
  Interventions: Other: Home Exercise Therapy

INTERVENTIONS:
Other: Manual Therapy — Various soft tissue and joint mobilizations, intramuscular stretches, trigger point treatments, and intraoral applications for the temporomandibular joint were performed in 15 randomly selected bruxism patients. Manual therapy was applied twice weekly over eight weeks, each session lasting approximately 45 minutes. Techniques included trigger point therapy, myofascial release, intraoral mobilizations to the masseter, medial and lateral pterygoid, and temporalis tendons, post-isometric relaxation for masticatory muscles, cervical traction, and suboccipital and cervical fascial release. The manual therapy procedure, which was applied in the supine position and lasted approximately 40 minutes for 8 weeks
  Arms: Manual Therapy Group
Other: Home Exercise Therapy — The exercise group consisted of 15 randomly selected bruxist individuals and aimed to reduce pain, decrease involuntary contractions of masticatory muscles, increase their nutrition, flexibility and coordination, and strengthen weak muscles with exercise therapy. The exercise program included Rocabado exercises, stretching of the platysma, masticatory and cervical muscles, resistance training (mouth opening, protrusion, and lateral mandibular movements), and postural exercises. Exercises were performed while sitting in a chair with back support in front of a mirror. Each exercise was repeated 10 times. The duration of each session was 25-30 minutes. repeat the home exercises three times a week for 8 weeks. Weekly phone calls were made to encourage compliance. In addition, a video explaining the exercises in detail was shared with all participants in the group in order to ensure that the exercises were not forgotten and to achieve accuracy and standardization among the participants.
  Arms: Exercise Group

SUMMARY:
Bruxism is a multifactorial condition that affects the masticatory muscles and often requires multidisciplinary management. This study aimed to investigate and compare the effects of manual therapy and home exercise on pain intensity, number of myofascial trigger points, temporomandibular joint (TMJ) and cervical mobility, head posture, muscle thickness, stiffness, and activity in individuals with bruxism.

Methods: Thirty individuals diagnosed with bruxism were randomly assigned to two intervention groups: the Home Exercise Group (HEG) and the Manual Therapy Group (MTG). All participants received education about bruxism. The HEG performed a supervised home-based exercise program three times per week for eight weeks, supported by instructional videos and weekly follow-up. The MTG received intraoral and extraoral manual therapy targeting the jaw and cervical regions twice a week over the same period. Pain intensity (Visual Analog Scale), trigger point count (palpation), TMJ mobility (ruler), head posture and cervical mobility (goniometer), muscle thickness and stiffness (ultrasound), and muscle activity (electromyography) were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer students aged between 18-25
* Answered "yes" to at least two of the six questions in the Bruxism questionnaire.

Is there anyone hear you grinding your teeth at night? Do you feel fatigue or pain in your jaw when you wake up in the morning? Do you feel pain in your teeth and gums when you wake up in the morning? Do you have a headache when you wake up in the morning? Do you notice that you grind your teeth during the day? Do you notice that you clench your teeth during the day?

-Having at least two clinical signs of bruxism Abnormal tooth wear on the occlusal surfaces of the teeth Abfraction Gingival recession and/or cervical defect Tongue indentations or damage to the inside of the cheek Tense facial and jaw muscles, muscle sensitivity, and masseteric hypertrophy upon bidigital palpation

Exclusion Criteria:

* Characterized by a neurological disease,
* Botulinum toxin injections into the masticatory muscles in the last year,
* Using antidepressant-type medications that will affect the central nervous system,
* Receiving occlusal splint treatment,
* Having more than two molar teeth missing in the posterior
* Individuals who cannot cooperate

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Pain Level | From baseline to the end of treatment at 8 weeks
  Visual analog scale (VAS) was used to assess the severity of pain related to bruxism. On a 10 cm long horizontal line, "0 (no pain)" was written at the beginning and "10 (most intense pain)" was written at the end and the patient was asked to mark the pain intensity they perceived at rest, active use and at night on the line. The pain intensity of the individual was recorded by measuring the distance marked on the line in millimeters. It has been reported that the Turkish version of the VAS is a valid and reliable measurement tool in the evaluation of musculoskeletal disorders
Cervical and Temporomandibular Joint Range of Motion (ROM) | From baseline to the end of the treatment at 8 weeks
  Cervical flexion, extension, lateral flexion, and rotation were measured using a universal goniometer. TMJ range of motion, including maximum mouth opening, protrusion, retrusion, and lateral excursions, was measured using a ruler.
Ultrasonographic Imaging | From baseline to the end of treatment at 8 weeks
  Ultrasound and elastography measurements were performed using the ACUSON S 2000 system (Siemens, Munich, Germany) by a single experienced radiologist. A 4-9 MHz linear transducer was used to measure the thickness and elasticity of the masseter, anterior temporalis, and SCM muscles both at rest and during maximal clenching, in a semi-recumbent position with head support. Measurements were recorded in millimeters
Electromyography (EMG) | From baseline to the end of treatment at 8 weeks
  Surface EMG recordings were obtained using an 8-channel EMG system (BioResearch Inc., Milwaukee, Wisconsin, USA). Self-adhesive disposable surface electrodes were placed bilaterally over the masseter, anterior temporalis, and SCM muscles, with a grounding electrode on the trapezius. Electrodes were aligned parallel to muscle fibers at the muscle belly. Measurements were conducted in a quiet, dimly lit room, with participants seated in the Frankfurt Horizontal Plane position. Participants were asked to clench their teeth three times and then relax. Each EMG recording lasted 10 seconds and was repeated twice. From each 10-second recording, three 2-second segments from the first 6 seconds were selected, and the average EMG activity was calculated.

SECONDARY OUTCOMES:
Trigger Point | From baseline to the end of treatment at 8 weeks
  While evaluating the trigger points in the masticatory and neck muscles, the tense muscle was palpated with a fingertip. Palpation was performed along the long axis of the tense muscle and the most sensitive point was determined. Sudden reaction or vocal response of the patient with light pressure applied to this point and the presence of reflected pain in a region distant from this region indicated the presence of a trigger point. Evaluation was performed in 14 muscles (masseter, temporalis, suprahyoid, sternocleidomastoid (SCM), scalene, and suboccipital muscles) and the muscles with trigger points and the total number of trigger points were recorded.
Presence and severity of Temporomandibular Joint Disorder (TMD) symptoms | From baseline to the end of treatment at 8 weeks
  It was examined with Fonseca Anamnestic Index (FAI). The Fonseca Anamnestic Index, a 10-question questionnaire designed to assess temporomandibular dysfunction (TMD), was administered. Responses included "No (0 points)," "Sometimes (5 points)," and "Yes (10 points)." The total score was calculated to quantify the severity of TMD. A high score means that the disorder is severe.
Bruxism | From baseline to the end of treatment at 8 weeks
  It was examined with Bruxism Questionnaire. According to the survey questions prepared by referencing the studies of Pintado, it was stated that individuals who answered "Yes" to at least two of the questions specified in the survey can be called bruxists. The total score range varies between 0-6. A high score means that the disorder is severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Health Services Vocational School, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Investgators can share the questionnaires and indexes used in the study
Supporting Information: Study Protocol